CLINICAL TRIAL: NCT07288229
Title: The Benefits of Wearable Device-Based Artificial Intelligence in Post-Discharge Management of Patients With Acute Myocardial Infarction
Brief Title: The Benefits of Wearable AI in Post-Discharge Management of AMI Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Zhiguo Zou, Doctor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EARLY-MYO Wearable AI
Record Dates: First submitted 2025-11-14; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Acute Myocardial Infarction; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The guideline-guided traditional management group (No Intervention): As the control group, wearable data will be collected but not shared with the participant and responding physician or used for clinical management during the study period. All management in the participants is based on updated clinical guidelines.
- The guideline-guided and wearable-assisted management group (Experimental): As the intervention group, in addition to clinical guidelines, wearable data and AI analytical results will be made available to both patients and their physicians. These insights will be discussed during follow-ups and used to support lifestyle modification, medication adjustment, and clinical decision-making.
  Interventions: Combination Product: Optimized Integrated Management Based on AI-Guided Wearable Data

INTERVENTIONS:
Combination Product: Optimized Integrated Management Based on AI-Guided Wearable Data — The collected data will be shared with both patients and their treating physicians during follow-up visits. Based on these insights, the clinical team will offer personalized recommendations regarding medication adjustment, lifestyle modification, diet optimization, and physical activity guidance.
  Arms: The guideline-guided and wearable-assisted management group

SUMMARY:
Myocardial infarction (MI) remains a major threat to human health. Although interventional treatment techniques have advanced rapidly, many patients still experience major adverse cardiovascular events (MACE) and require hospital readmission after discharge. Artificial intelligence (AI) based on wearable device data has shown great potential in the diagnosis and management of cardiovascular diseases.

This study aims to explore the clinical value of wearable device-based data analysis and AI-driven risk stratification models in post-discharge management of acute myocardial infarction (AMI) patients.

DETAILED DESCRIPTION:
This prospective, open-label, randomized controlled study aims to evaluate the clinical benefits of wearable device-based AI risk models in post-discharge management of AMI patients. A total of 200 patients who have undergone PCI and provided informed consent will be enrolled, including those with both preserved and reduced left ventricular ejection fraction (LVEF).

Participants will be randomly assigned to either the control group or the intervention group in a 1:1 ratio. All patients will be equipped with a wearable smartwatch and continuously monitored for 3 months after discharge. Data collected will include physiological signals, sleep and activity parameters. In both groups, patients will receive weekly telephone follow-ups and monthly office visits to record symptoms, medication use, and adverse events.

In the intervention group, wearable data and AI analytical results will be made available to both patients and their physicians. These insights will be discussed during follow-ups and used to support lifestyle modification, medication adjustment, and clinical decision-making. In the control group, AI data will be collected but not shared or used for clinical management during the study period.

The primary study endpoint is the time to first unplanned hospital readmission within 3 months, including readmissions due to chest pain, heart failure, arrhythmia, recurrent myocardial infarction, or death. The secondary endpoints include: Change in Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) score from baseline to 3 months; change in left ventricular ejection fraction (LVEF) measured by echocardiography between baseline and 3 months.

The investigators hypothesize that AI-assisted, wearable-based monitoring and feedback will improve early detection of adverse cardiovascular events, reduce unplanned hospitalizations, increase LVEF in patients with reduced LVEF at discharge, and enhance quality of life compared with standard post-discharge care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years.
* Confirmed diagnosis of acute myocardial infarction (AMI), including both ST-segment elevation myocardial infarction (STEMI) and non-ST-segment elevation myocardial infarction (NSTEMI).
* Underwent successful percutaneous coronary intervention (PCI) during index hospitalization.
* Hemodynamically stable at the time of hospital discharge.
* Willing and able to wear a smartwatch continuously for the study period.
* Compatible with the data collection application and have stable internet access.

Exclusion Criteria:

* Planned staged or elective PCI or any coronary revascularization scheduled within 3 months after discharge.
* Unable to tolerate or contraindicated for wearing metal or electronic monitoring devices.
* Pregnant or breastfeeding women.
* Residence in an area without stable network connectivity or inability to use a smartphone for data upload and communication.
* Severe comorbidities that limit 3-month survival or follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to First Unplanned Re-hospitalization event | From the date of hospital discharge to 3 months post-discharge (90 days).
  The primary study endpoint is the time to first unplanned hospital readmission within 3 months, including readmissions due to chest pain, heart failure, arrhythmia, recurrent myocardial infarction, or death.

SECONDARY OUTCOMES:
Change in LVEF | At baseline and at 3 months post-discharge
  LVEF will be assessed by transthoracic echocardiography at discharge (baseline) and at 3 months post-discharge follow-up. The change in LVEF will be calculated as the difference between the two measurements.
Change in the score of Kansas City Cardiomyopathy Questionnaire-12 | At baseline and at 3 months post-discharge.
  The KCCQ-12, a validated patient-reported outcome measure, will be administered during the index hospitalization (prior to discharge) and again at 3 months post-discharge follow-up.